CLINICAL TRIAL: NCT02183467
Title: Assessment of the Effect of 5 mg and 100 mg of BI 1356 as Single Dose on the QT Interval in Healthy Female and Male Subjects. A Randomised, Placebo Controlled, Double-blind, Four-way Crossover Study With Moxifloxacin as Positive Control
Brief Title: Effect of BI 1356 as Single Dose on the QT Interval in Healthy Female and Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.32
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Moxifloxacin

ARMS (4):
- BI 1356, low dose (Experimental)
  Interventions: Drug: BI 1356, low dose
- BI 1356, high dose (Experimental)
  Interventions: Drug: BI 1356, high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Moxifloxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: BI 1356, low dose
  Arms: BI 1356, low dose
Drug: BI 1356, high dose
  Arms: BI 1356, high dose
Drug: Placebo
  Arms: Placebo
Drug: Moxifloxacin
  Other Names: Avalox®
  Arms: Moxifloxacin

SUMMARY:
Assessment of the effect of BI 1356 or Placebo on prolongation of the QT interval

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females, 21 to 50 years of age
* Body mass index (BMI) ranging from 18.5 to 29.9 kg/m2
* Signed written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than ten half-lives of the respective drug before enrolment in the study or during the study
* Use of any drugs which might influence the results of the trial up to 7 days prior to enrolment in the study or during the study
* Participation in another trial with an investigational drug (≤ 60 days prior to administration or during the trial)
* Heavy smoker (> 10 cigarettes or > 3 cigars of > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (> 60 g/day)
* Drug abuse
* Blood donation (≥ 100 mL within four weeks prior to administration or during the trial)
* Any deviation of a laboratory value that is considered to be of clinical relevance
* Excessive physical activities within the last week before the trial or during the trial
* Hypersensitivity to Moxifloxacin or related drugs of these classes
* Supine blood pressure at screening of systolic < 100 mmHg and diastolic < 60 mmHg
* Heart rate at screening of > 80 bpm or < 40 bpm
* Any screening ECG value outside of the reference range of clinical relevance including, but not limited to PR interval > 220 ms, QRS interval > 115 ms, QTcB or QTcF > 450 ms, or QT (uncorrected) > 470 ms
* Subjects involved in passenger transport or operation of dangerous machines

For Female subjects:

* Pregnancy or positive pregnancy test, or planning to become pregnant during the study or within 1 month of study completion Pregnancy
* No adequate contraception during the study and until 1 month of study completion, i.e. implants, injectables, combined oral contraceptives, IUD [intrauterine device], sexual abstinence (for at least 1 month prior to enrolment), vasectomised partner (vasectomy performed at least 1 year prior to enrolment), or surgical sterilisation (incl. hysterectomy). Females, who have not a vasectomised partner, are not sexually abstinent or surgically sterile will be asked to additionally use barrier contraception methods (e.g. condom, diaphragm with spermicide)
* Lactation period

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2008-01; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline of the QTcI interval (individually heart rate-corrected QT interval length) | Pre-dose and 1 to 4 hours following administration

SECONDARY OUTCOMES:
Mean of the QTcI change from baseline of all electrocardiograms (ECGs) taken from 1 hour to 24 hours after dosing | up to 24 hours following administration
Change from mean baseline of the QTcI at any point in time between 1 and 24 hours after dosing | up to 24 hours following administration